CLINICAL TRIAL: NCT06480656
Title: Eccentric Cycling Exercise During Pulmonary Rehabilitation in Pulmonary Vascular Disease
Brief Title: Eccentric Cycling Exercise During Pulmonary Rehabilitation Pulmonary Vascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Silvia Ulrich Somaini, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EccRehab
Record Dates: First submitted 2024-05-31; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Eccentric Cycling Exercise
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric cycling exercise (Experimental)
  Interventions: Procedure: Rehabilitation with eccentric cycling exercise
- Concentric cycling exercise (Active Comparator)
  Interventions: Procedure: normal rehabilitation

INTERVENTIONS:
Procedure: Rehabilitation with eccentric cycling exercise — Instead of normal cycling, patients will exercise on the eccentric bike.
  Arms: Eccentric cycling exercise
Procedure: normal rehabilitation — Normal rehabilitation will be conducted
  Arms: Concentric cycling exercise

SUMMARY:
Eccentric cycling allows high intensities with low metabolic costs. Therefore the aim of this project is to investigate whether ECC improves exercise capacity and possibly hemodynamics during prolonged rehabilitation programs in patients with PVD

DETAILED DESCRIPTION:
Eccentric cycling exercise (ECC) allows training at low metabolic costs and may therefore be valuable for patients with pulmonary vascular disease (PVD). For these patients, regular exercise training has an evidence level 1A recommendation in the current guidelines. Exercise training during longer and regular periods provides chronic adaptation, for which ECC was recently found to have a greater effectiveness than CON by increasing muscle strength, hypertrophy, six-minute walking distance and furthermore, by increasing maximum oxygen uptake (V'O2max) especially in patients with chronic obstructive pulmonary disease (COPD), chronic left heart failure or coronary heart disease.

Furthermore, the investigators conducted an RCT in which the investigators exposed patients with PVD to ECC and concluded that ECC is a feasible and well-tolerated exercise modality for PVD patients with severely lower O2 demand and load to the right ventricle.

Therefore the aim of this project is to investigate whether ECC improves exercise capacity and possibly hemodynamics during prolonged rehabilitation programs in patients with PVD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PVD, either PAH or CTEPH according to recent guidelines
* Stable medication for at least 1 month
* Age 18 to 85 years
* No resting hypoxemia (PaO2 >7.3kPa)

Exclusion Criteria:

* Any co-morbidity that limits the patient to participate the full rehabilitation
* Enrollments in other trials with active treatments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
peak exercise capacity | 3 weeks

SECONDARY OUTCOMES:
Peak oxygen uptake | 3 weeks
  Assesses during exercise until exhaustion using an incremental exercise protocol
ventilatory equivalent for CO2 | 3 weeks
Finger pulseoximetry | 3 weeks
  Arterial oxygen saturation will be assessed by finger clip Infrared spectroscopy
6 minute walk distance | 3 weeks
systolic pulmonary artery pressure | 3 weeks
total pulmonary resistance | 3 weeks
ventricular - pulmonary arterial coupling | 3 weeks
cardiac output | 3 weeks
  will be assessed by echocardiography using the pulse-wave doppler technique at the left ventricular outflow tract durig systole.
Arterial partial pressure for oxygen | 3 weeks
  Arterial blood gas analyses, taken from the radial artery and analysed by radiometer
Arterial partial pressure for carbon dioxide | 3 weeks
  Arterial blood gas analyses, taken from the radial artery and analysed by radiometer
Arterial oxygen saturation | 3 weeks
  Arterial blood gas analyses, taken from the radial artery and analysed by radiometer
Arterial lactate concentration | 3 weeks
  Arterial blood gas analyses, taken from the radial artery and analysed by radiometer
Borg CR 10 for perceived dyspnea | 3 weeks
Borg CR 10 for perceived leg fatigue | 3 weeks
Visual analogue scale generell well being | 3 weeks
Visual analogue scale dyspnea | 3 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Rehabilitation clinic Barmelweid, Erlinsbach
  - University Hospital Zurich, Pneumology, Zurich

IPD SHARING:
Plan to Share IPD: Undecided